CLINICAL TRIAL: NCT05628857
Title: A Study to Evaluate the Efficacy, Safety and Pharmacokinetics of RC108 for Injection in the Treatment of Patients With c-Met-positiveAdvanced Digestive System Malignant Tumor
Brief Title: A Study of RC108-ADC in Subjects With Advanced Digestive System Malignant Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC108-C002
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-04

CONDITIONS: Digestive Cancer
Keywords: Digestive Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): gastric cancer patients
  Interventions: Drug: RC108
- cohort 2 (Experimental): colorectal cancer patients
  Interventions: Drug: RC108
- cohort 3 (Experimental): liver cancer patients
  Interventions: Drug: RC108
- cohort 4 (Experimental): other digestive system malignancies, including esophageal cancer, pancreatic cancer, gallbladder cancer, etc.
  Interventions: Drug: RC108

INTERVENTIONS:
Drug: RC108 — RC108 is comprised of an antibody component conjoined to a drug component in a lyophilized powder, which is made into solution for intravenous administration.

SUMMARY:
A multi-center, open-label, study designed to evaluate the preliminary efficacy, safety and pharmacokinetics of RC108 in patients with c-Me-positive advanced digestive system malignancies.

DETAILED DESCRIPTION:
The primary purpose of this trial is to evaluate the preliminary efficacy, safety and efficacy of RC108 in patients with c-Me positive advanced gastrointestinal malignancies such as gastric, colorectal, esophageal, hepatic, pancreatic and bile duct cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary agreement to provide written informed consent.
2. Male or female, aged between 18 to 75 years.
3. Predicted survival for ≥ 12 weeks. Diagnosed with histologically or cytologically confirmed locally advanced or metastatic Digestive System Malignant Tumor.
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
5. All female subjects will be considered to be of child-bearing potential unless they are postmenopausal, or have been sterilized surgically. Female subjects of child-bearing potential must agree to use two forms of highly effective contraception. Male subjects and their female partner who are of child-bearing potential must agree to use two forms of highly effective contraception.
6. Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

   Adequate organ function, evidenced by the following laboratory result Participant has adequate bone marrow, renal, and hepatic function.
7. bone marrow function: Hemoglobin ≥ 9g/dL; Absolute neutrophil count ≥ 1.5×10^9 /L Platelets ≥ 100×10^9 /L.
8. hepatic function: Total bilirubin ≤ 1.5× ULN; AST and ALT ≤ 2.5×ULN and ≤ 5 x ULN with hepatic metastasis
9. renal, and hepatic function: Serum creatinine ≤1.5×ULN.
10. Cardiac ejection fraction ≥ 50%. Median QTc < 450 ms.
11. c-Met positive as confirmed by the central laboratory.
12. Measurable lesion according to RECIST 1.1.

Exclusion Criteria:

1. Known hypersensitivity to the components of RC108-ADC.
2. Toxicity of previous anti-tumor treatment not recovered to CTCAE (v5.0) Grade 0-1 (with exception of Grade 2 alopecia).
3. Uncontrolled pericardial effusion or cardiac tamponade, or pleural or abdominal effusion with clinical symptoms.
4. History of receiving any anti-cancer drug/biologic treatment within 4 weeks prior to trial treatment.
5. History of major surgery within 4 weeks of planned start of trial treatment.
6. Has received a live virus vaccine within 4 weeks of planned start of trial treatment.
7. Currently known active infection with HIV or tuberculosis.
8. Diagnosed with HBsAg, HBcAb positive and HBV DNA copy positive, or HCVAb positive.
9. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
10. History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
11. Known central nervous system metastases.
12. Uncontrolled hypertension, diabetes, pulmonary fibrosis, acute lung disease, Interstitial lung disease, or liver cirrhosis;
13. Pregnancy or lactation.
14. Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 Months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
DCR | Up to 24 Months
  The disease control rate is the proportion of those subjects with complete response, partial response, or stable disease, as defined by Response Evaluation Criteria in Solid Tumors Criteria (RECIST 1.1)
Adverse Events | Up to 24 Months
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
DOR | Up to 24 Months
  DOR is defined as the time from the participant's initial objective response to study drug therapy to disease progression or death, whichever occurs first.
TTP | Up to 24 Months
  Time to progression will be measured from the first day of study drug until progression.
PFS | Up to 24 Months
  PFS time is defined as the time from the participant's first dose of RC108 to either the participant's disease progression or death, whichever occurs first.
OS | Up to 5 years
  Duration from date of sub-study registration (or date of screening/pre-screening registration if patient never enrolls in a sub-study) to date of death due to any cause.
Area under the curve (AUC) from time zero to the last measurable concentration AUC (0-t) | Up to 24 Months
  Area under the curve (AUC) from time zero to the last measurable concentration AUC (0-t)
Maximum observed plasma concentration (Cmax) | Up to 24 Months
  Maximum observed plasma concentration (Cmax)
Time to Cmax (Tmax) | Up to 24 Months
  Time to Cmax (Tmax).
Terminal elimination half life | Up to 24 Months
  Terminal elimination half life.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Fang, Ph.D, Study Director — RemeGen Co., Ltd.
Locations (1):
- Beijing Cancer Hopspital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No